CLINICAL TRIAL: NCT02671461
Title: A Phase 2, Placebo Controlled, Randomized, Double-Blind, Parallel-Arm Study to Evaluate Efficacy and Safety of BMS- 986141 For the Prevention of Recurrent Brain Infarction in Subjects Receiving Acetylsalicylic Acid (ASA) Following Acute Ischemic Stroke or Transient Ischemic Attack
Brief Title: Safety and Efficacy Study of a Protease Activated Receptor-4 Antagonist Being Tested to Reduce the Chances of Having Additional Strokes or "Mini Strokes"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV006-004
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — BMS-986141; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMS-986141 0.8mg (Experimental): BMS-986141 0.8mg orally (tablets) and Aspirin (ASA) 75 to 162 mg orally (tablets)
  Interventions: Drug: BMS-986141; Drug: Aspirin
- BMS-986141 4.8mg (Experimental): BMS-986141 4.8mg orally (tablets) and ASA 75 to 162 mg orally (tablets)
  Interventions: Drug: BMS-986141; Drug: Aspirin
- Placebo (Placebo Comparator): Placebo orally (tablets) and ASA 75 to 162 mg orally (tablets)
  Interventions: Drug: Aspirin; Other: Placebo

INTERVENTIONS:
Drug: BMS-986141
  Arms: BMS-986141 0.8mg; BMS-986141 4.8mg
Drug: Aspirin
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BMS-986141 is effective in reducing the recurrence of stroke in people who recently had a stroke, or a transient ischemic attack (known as a TIA or "mini stroke") and are receiving acetylsalicylic acid (also known as aspirin or ASA) to treat the stroke or TIA.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female, age 18 or older
* Must have had a very recent stroke or transient ischemic attack ("mini stroke") that can be confirmed by the study doctor
* Able to be assigned to a study group no later than 48 hours after the stroke occurred
* Has an image of the brain that confirms that the stroke was not caused by hemorrhage or other reason that could explain symptoms

Exclusion Criteria:

* A suspicion by the study doctor that the transient ischemic attack or stroke was caused by a blood clot that formed in the heart; examples of this include history of an abnormal heart rhythm known as atrial fibrillation or a ventricular aneurysm or defect of the heart.
* Any condition requiring treatment with an anticoagulant
* History of intracranial hemorrhage ("bleeding in the brain")
* Gastrointestinal ("stomach or intestinal") bleeding in the last 3 months that required treatment
* Planned or anticipated invasive surgery or procedure during the study
* Unable to tolerate MRI procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (27):
  - Banner University Medical Ctr, Phoenix, Arizona
  - Hoag Memorial Hospital, Newport Beach, California
  - Local Institution, Newark, Delaware
  - University Of Florida, Gainesville, Florida
  - University Of Florida Hsc/Jacksonville, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - University Of Louisville, Louisville, Kentucky
  - Local Institution, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - St. Lukes Marion Bloch Neuroscience Institute, Kansas City, Missouri
  - Advanced Neurology Specialists, Great Falls, Montana
  - Local Institution, Omaha, Nebraska
  - JFK Medical Center, Edison, New Jersey
  - Local Institution, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Guilford Medical Associates, Pa, Greensboro, North Carolina
  - Providence Portland Med Ctr, Portland, Oregon
  - Providence St Vincent Medical Center, Portland, Oregon
  - Oregon Health Science Univ, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - Local Institution, Memphis, Tennessee
  - West Virginia University, Morgantown, West Virginia
- Japan (6):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Sendai, Miyagi
  - Local Institution, Hidaka-shi, Saitama
  - Local Institution, Fukuoka

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were enrolled; 15 were randomized; 14 were treated. 1 participant was not randomized because the interactive voice response system did not work at the time of enrollment
Groups:
- Placebo: Matching placebo was taken once daily. Administration was exactly the same as for BMS-986141
- BMS-986141 0.8 mg: BMS-986141 0.8 mg QD for up to 28 days
- BMS-986141 4.8 mg: BMS-986141 4.8 mg QD for up to 28 days
Period: Treatment
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Started | 3 | 5 | 7
Completed | 1 | 2 | 2
Not Completed | 2 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Administrative Reason by Sponsor | 1 | 3 | 4
Not completed — Randomized, not treated | 1 | 0 | 0
Period: Follow-up
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Started | 2 | 5 | 7
Completed | 1 | 4 | 6
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Administrative Reason by Sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg | Total
Number analyzed (Participants) | 3 | 5 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants
  years | 63.3 (9.2) | 64.8 (12.2) | 66.7 (7.6) | 65.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized participants
  Participants
    Female | 1 | 1 | 3 | 5
    Male | 2 | 4 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 3 | 5 | 7 | 15
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 1 | 3
    White | 3 | 3 | 5 | 11
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Symptomatic Ischemic Stroke by Day 28 and Unrecognized Brain Infarction Assessed by MRI at Day 28
Description: The incidence of a composite of symptomatic ischemic stroke by Day 28 and unrecognized brain infarction assessed by MRI at Day 28 was to be reported by arm in all treated participants.
Time Frame: 28 Days
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Composite of Adjudicated Major Bleeding and Adjudicated Clinically Relevant Non-major (CRNM) Bleeding During the Treatment Period
Description: The percentage of participants with composite of major bleeding and CRNM bleeding was to be reported. Point estimates and 95% CIs for event rates were to be presented by treatment, together with point estimates and 95% CIs for the difference of event rates between each BMS-986141 arm and placebo.
Time Frame: Up to 90 days
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Major Adverse Cardiovascular Events (MACE)
Description: MACE was defined as a composite of adjudicated recurrent stroke, myocardial infarction, or cardiovascular death. The percentage of treated participants experiencing these events at Day 90 was to be reported by arm.
Time Frame: 90 days
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Adjudicated Symptomatic Recurrent Stroke (Including Fatal and Non-fatal)
Description: The percentage of participants with adjudicated symptomatic recurrent stroke at Day 28 was to be reported by arm for all treated participants.
Time Frame: Day 28
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Composite of Unrecognized Brain Infarction Assessed by MRI at Day 28 and MACE at Day 90
Description: The percentage of participants with unrecognized brain infarction at Day 28 and MACE at Day 90 was to be reported by arm for all treated participants.
Time Frame: Day 90
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Composite of Adjudicated Recurrent Ischemic Stroke, Myocardial Infarction, or Cardiovascular Death
Description: The percentage of treated participants with composite of adjudicated recurrent ischemic stroke, myocardial infarction, or cardiovascular death was reported by arm.
Time Frame: Day 90
Population: Insufficient data available to perform analysis due to study termination
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose until 30 days following last dose (assessed up to March 2017, approximately 6 months)
Arm/Group | Placebo | BMS-986141 0.8 mg | BMS-986141 4.8 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 1/7
Other Adverse Events (participants affected / at risk) | 0/3 | 4/5 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | BMS-986141 0.8 mg (N=5) | BMS-986141 4.8 mg (N=7)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | BMS-986141 0.8 mg (N=5) | BMS-986141 4.8 mg (N=7)
Blood Potassium Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Pruritis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Micturation Urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT02671461/SAP_000.pdf
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02671461/Prot_001.pdf